CLINICAL TRIAL: NCT03505645
Title: Surgical Techniques in Arthroplasty of the Knee (STArK) 1 Trial: Periarticular Infiltration Versus Intra-articular Injection for Postoperative Analgesia in Primary Total Knee Arthroplasty: a Randomised Double Blind Controlled Trial
Brief Title: Surgical Techniques in Arthroplasty of the Knee (STArK) 1 Trial
Acronym: STArK1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chloe Scott (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor-Investigator, Chloe Scott, Consultant Orthopaedic Surgeon, Royal Infirmary of Edinburgh
Organization: Royal Infirmary of Edinburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 241807
Record Dates: First submitted 2018-04-04; First posted 2018-04-23 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group 1: Periarticular infiltration (Active Comparator): Patients undergoing total knee replacement who are randomised to Treatment Group 1.
  Interventions: Procedure: Periarticular infiltration
- Treatment Group 2: Intra-articular infiltration (Active Comparator): Patients undergoing total knee replacement who are randomised to Treatment Group 2.
  Interventions: Procedure: Intra-articular infiltration

INTERVENTIONS:
Procedure: Periarticular infiltration — The injection will consist of the same drugs for all patients: 150mg levobupivacaine 0.25%, 10mg morphine; and 30mg ketorolac made up to a volume of 150ml with saline.
  The difference between treatment groups is how the multimodal injection is administered: either by periarticular infiltration around the knee, or by simple intra-articular injection after the knee joint capsule has been closed.
  Treatment group 1: Periarticular infiltration
  Intra-operatively after bone cuts have been made and prior to implant cementation, the multimodal injection will be infiltrated around the knee at 6 specific sites:
  1. Medial femoral condyle periosteum
  2. Medial gutter
  3. Lateral femoral condyle periosteum
  4. Lateral gutter
  5. Posteromedial capsule
  6. Posterolateral capsule
  Arms: Treatment group 1: Periarticular infiltration
Procedure: Intra-articular infiltration — The injection will consist of the same drugs for all patients: 150mg levobupivacaine 0.25%, 10mg morphine; and 30mg ketorolac made up to a volume of 150ml with saline.
  The difference between treatment groups is how the multimodal injection is administered: either by periarticular infiltration around the knee, or by simple intra-articular injection after the knee joint capsule has been closed.
  After implant cementation and watertight joint capsular closure, the multimodal injection will be injected intra-articularly through the closed capsule.
  Arms: Treatment Group 2: Intra-articular infiltration

SUMMARY:
Study Background Osteoarthritis of the knee is a common degenerative musculoskeletal condition which affects nearly five million people in the United Kingdom. Some patients will require total knee replacement surgery if their symptoms of pain and disability are not controlled adequately by so-called 'conservative' measures such as weight-loss, activity modification and analgesic (pain-killer) medication.

Over the past ten years our understanding of pain-relief strategies during total knee replacement, often termed 'Enhanced Recovery' principles, has helped improve patient care and reduced length of hospital admission. 'Enhanced Recovery' principles recommend the use of analgesic medications which can be delivered in a variety of ways e.g. tablets and injections. This is termed 'multi-modal' analgesia.

Prior to total knee replacement, the patient will receive an injection around the nerves in the spine (regional anaesthesia) which numbs the patient from the waist down and allows the surgeon to perform the operation in a safe and pain-free manner. During the operation, surgeons often choose to deliver extra local anaesthetic to prolong the degree of pain-relief in the immediate post-operative period. This can enable patients to mobilise early and is associated with greater long-term satisfaction.

There are two main methods of delivering this extra form of pain-relief during the operation. Peri-articular injection involves multiple injections of local anaesthetic into the soft-tissues surround the knee. In contrast, Intra-articular injection involves a single injection directly into the knee joint once the operation is finished. Currently, there is no clear evidence available to Orthopaedic surgeons to inform us which technique is better at providing pain relief for patients undergoing total knee replacement surgery.

All patients undergoing total knee replacement surgery for osteoarthritis of the knee will be invited to participate in this study. We intend to recruit a total of 120 patients. During the patient's total knee replacement surgery, they shall receive an injection of local anaesthetic around the soft-tissues of the knee (Peri-Articular Injection) or directly into the knee joint itself (Intra-Articular Injection). The decision regarding which treatment they receive is decided entirely by randomisation.

Following the operation, a member of the research team will assess the patient on the ward to collect information regarding levels of pain and overall satisfaction. The type of injection received shall be kept secret from both the patient and the member of the research team collecting the post-operative pain scores.

After the patient has been safely discharged from hospital, we intend to follow-up all participants for one year. This will involve routine clinic appointments at six weeks and twelve months following surgery. This will involve review and clinical examination by a member of the orthopaedic team who have treated the patient whilst in hospital and/or a member of the research team.

In addition, all patients will be asked to complete a questionnaire at twelve months regarding their level of function and pain. These questionnaires have been used widely in the medical literature and have a strong evidence base for their use.

What is the aim of this study? The aim of this study is compare the amount of pain relief provided by two different methods of local anaesthetic injection techniques used in total knee replacement surgery. In addition, we would like to know if this influences the patient's immediate and long-term recovery after surgery.

DETAILED DESCRIPTION:
The aim of this study is compare the amount of post-operative pain relief provided by two different methods of local anaesthetic injection techniques used in total knee replacement surgery.

'Enhanced Recovery After Surgery' protocols has significantly shortened recovery-time and length of hospital admission after total knee replacement (TKR). A major factor in this improvement has been the incorporation of multi- modal therapies which deliver adequate pain relief, limit post-operative nausea and enable early mobilisation.

Peripheral nerve blocks are performed by the anaesthetist immediately prior to surgery. This involves injecting local anaesthetic around the nerves which supply sensation around the knee. Injecting directly into the nerve can damage it and lead to significant disability. For this reason peripheral nerve blocks are often performed under ultrasound guidance. This can be time-consuming and does not negate the risk of nerve injury.

Peri-articular infiltration is performed during the operation by the surgeon. In the knee this involves injecting a solution of local anaesthetic into multiple specified soft-tissue and bony regions around the knee. It is performed blind without ultrasound guidance and also carries risk of nerve injury.

Intra-articular injections involve the surgeon injecting local anaesthetic solution into the knee joint itself. During TKR, this can be performed after closure of the joint capsule immediately prior to skin closure. This avoids risks to nerves and arteries as it is placed into the large knee joint, and not blindly around the joint capsule. In addition, it is simple to perform and less time-consuming than peri-articular infiltration.

Randomised controlled trials have previously compared femoral (peripheral) nerve blocks to periarticular infiltration, periarticular infiltration with and without posterior capsule infiltration, and periarticular infiltration to the front versus the back of the knee. However, to our knowledge the technique of intra-articular injection has not been compared to peri- articular infiltration for immediate post-operative analgesia following total knee arthroplasty

Study Design A double-blind randomised controlled trial (RCT) will be conducted in a single hospital, with four Consultant Knee Surgeons recruiting patients. It is anticipated from a previous RCT performed at the same centre, that recruitment be completed within 2 years.

Participants All patients undergoing primary total knee replacement for osteoarthritis under the care of 4 Consultant Orthopaedic Surgeons at the Royal Infirmary of Edinburgh will be assessed for eligibility for study enrolment.

All patients will receive trial information (patient information sheet) when they are placed on the waiting list for TKR. Patients currently wait 12 weeks for surgery. When patients are reviewed at a pre-assessment clinic 2-4 weeks prior surgery, those who fulfil the inclusion criteria will have the trial explained in full by the research team, supervised by the lead investigator Ms Chloe Scott, and will decide whether they wish to be involved. Informed consent will be obtained at this stage. Patients will then have 2-4 weeks before surgery to opt out of the study if they wish.

Power Calculation Audit of 10 TKR patients measuring VAS pain scores at 6 and 24 hours has demonstrated a standard deviation of 2.14 points. The minimum clinically important difference (MCID) for this score is 12mm (1.2 points). Assuming approximate normality for the VAS, primary outcome data on 102 patients (51 in each arm) will be required for 80% power at 5% significance. Allowing for a dropout rate of 10%, 120 patients will be recruited.

Randomization A total of 120 participants will be randomized in a 1:1 ratio to either Treatment Group 1 (periarticular infiltration) or Treatment Group 2 (intraarticular injection) using the sealed opaque envelope randomization technique. This will be performed after spinal anaesthetic has been administered before surgery commences.

Baseline information All patients will be initially evaluated with a complete history and physical examination. For all patients entering the study the following baseline information will be recorded: Age, sex, BMI, Kellgren-Lawrence grade of osteoarthritis, preoperative analgesia regime, length of knee pain duration, employment status, and postcode. Baseline VAS Pain scores, Oxford Knee Scores and EQ-5D scores will be collected as is routine for all of our arthroplasty patients.

Peri-operative Protocol All patients will be admitted on the day of surgery and undergo a standardised enhanced recovery anaesthetic protocol including spinal anaesthetic (with no intrathecal diamorphine) and no peripheral nerve blocks (femoral, sciatic or adductor canal).

All patients will undergo a cemented Triathlon (Stryker, Mahwah, NJ, USA) cruciate retaining TKR.

All patients will be prescribed standardised post-operative analgesia including Oxycodone MR 15mg twice daily for 4 doses with stepdown to weaker opiate, usually Cocodamol 30/500 2 tabs 4 times per day, Oxycodone IR 5-10mg prn for breakthrough pain.

Patients will be placed first or second on the operating list to enable VAS pain scores to be collected at the assigned times.

Multimodal injection The injection will consist of the same drugs for all patients: 150mg levobupivacaine 0.25%, 10mg morphine; and 30mg ketorolac made up to a volume of 150ml with saline.

The difference between treatment groups is how the multimodal injection is administered: either by periarticular infiltration around the knee, or by simple intra-articular injection after the knee joint capsule has been closed.

Treatment group 1: Periarticular infiltration

Intra-operatively after bone cuts have been made and prior to implant cementation, the multimodal injection will be infiltrated around the knee at 6 specific sites:

1. Medial femoral condyle periosteum
2. Medial gutter
3. Lateral femoral condyle periosteum
4. Lateral gutter
5. Posteromedial capsule
6. Posterolateral capsule

Treatment Group 2: Intra-articular infiltration After implant cementation and watertight joint capsular closure, the multimodal injection will be injected intra-articularly through the closed capsule.

Post-operative protocol and Follow-up Postoperatively patients will complete a VAS pain score at 6, 12 24 and 48 hours postoperatively with research staff blinded to the infiltration technique employed. All analgesia required in the first 24 hours will be recorded and an opiate equivalency dose calculator used to determine opiate intake (Joint Formulary Committee 2016). At 48 hours, in addition to recording a VAS pain score, patients will be asked how satisfied they were with their pain relief as scored on a 5 point Likert score from very satisfied to very dissatisfied.

Patients will then undergo routine postoperative management with review by arthroplasty practitioners blinded to their treatment arm at 6 weeks where they will be examined and will be asked to complete an adverse events questionnaire.

Patient reported outcomes including Oxford Knee Scores and EQ-5D scores will be collected as standard at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee osteoarthritis requiring Total Knee Replacement surgery
* Planned for cruciate retaining prosthesis without patella resurfacing
* Patient is able to give informed consent
* Patient resides locally and will be available for follow up

Exclusion Criteria:

* Inflammatory arthropathy
* Preoperative morphine based analgesia
* Renal insufficiency (GFR<30)
* Allergy to study drugs
* Spinal anaesthetic not possible
* Neurological disorder affecting the lower limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in pain levels during first 48 hours after surgery. | Pre-operative baseline and then re-checked at intervals in post-operative period 6, 12, 24 and 48 hours
  The Visual Analogue Score (VAS) for pain is a well recognised and validated measure of postoperative pain and has been used as a primary outcome measure on other studies comparing analgesic methods at Total Knee Replacement

SECONDARY OUTCOMES:
Opiate use first 24 hours | 24 hours
  We will record amount of regular and as required opiates required for pain relief in initial recovery period.
Length of hospital stay | Through study completion, at 12 months post-operation.
  Measurement of duration of hospital admission following elective total knee replacement.
Patient Satisfaction | Through study completion, at 12 months post-operation.
  Patients will be asked to rate their level of satisfaction with operation and recovery using Likert scale.
Change in Oxford Knee Score at 12 months after surgery. | 12 months
  The Oxford Knee Score (OKS) is a validated measure of pain and function following total knee replacement. The OKS is comprised of 12 questions which can be scored from 0 to 4 (with 0 being the worst outcome and 4 being the best outcome). The scores are then summed up to produce an overall score running from 0 (worst possible) to 48 (best possible). The OKS has sub-scales based on 'Functional Components' (questions 2, 3, 7, 11, 12) and 'Pain Components' (Questions 1, 4, 5, 6, 8, 9, 10). A raw score is created for each sub-scale based on the 0-4 scoring system. To enable easier interpretation, each sub-scale is standardised to a range from 0 (worst possible) to 100 (best possible). This is done by multiplying the 'Functional Component' raw score by 5 and 'Pain Component' score by 3.57. We intend to record and report the change in Pre-operative and 12 months post-operative OKS using the total score and also providing data on the Pain and Functional Component scores.

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Scott, FRCSEd, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No patient identifiable data shall be available to anyone other than the trial researchers.